CLINICAL TRIAL: NCT02467686
Title: Effects of Cimicifuga Racemosa L. Nutt Sexuality of Women With Breast Cancer Using Tamoxifen or Aromatase Inhibitor
Brief Title: Breast Cancer, Sexuality and Black Cohosh
Acronym: Cimicifuga
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Irmandade da Santa Casa de Misericordia de Sao Paulo (Other)
Responsible Party: Principal Investigator, Carolina Furtado Macruz, Doctor, Irmandade da Santa Casa de Misericordia de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 349441
Record Dates: First submitted 2015-03-04; First posted 2015-06-10 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Sexuality
MeSH Terms: conditions — Sexuality | interventions — Surveys and Questionnaires; black cohosh root extract; Tamoxifen; exemestane; Aromatase Inhibitors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cimicifuga racemosa (Active Comparator): The other group will have 30 patients receiving tamoxifen 20 mg orally daily or exemestane (aromatase inhibitor) 25 mg orally once daily after a meal and will start with 2 tablets per day of dry extract of Cimicifuga racemosa.
  Each tablet contains 20 mg of dry extract of Cimicifuga racemosa standardized between 1 mg and 1.25 mg of triterpene glycosides expressed in 26-deoxyactein. Will be guided 1 tablet 12/12 hours for 6 months.
  WHOQOL questionnaire (The World Health Organization Quality of life)application for evaluation at the first visit, 3-month and 6-month follow-up.
  FSFI questionnaire application for evaluation of sexual function at the first visit, 3-month and 6-month follow-up.
  Interventions: Behavioral: WHOQOL questionnaire; Behavioral: FSFI questionnaire; Behavioral: kupperman scale; Drug: Cimicifuga racemosa; Drug: tamoxifen; Drug: exemestane
- Control (Placebo Comparator): Control group will have 30 patients receiving tamoxifen 20 mg orally daily or exemestane (aromatase inhibitor) 25 mg orally once daily after a meal . They will be followed for 6 months and answer Kupperman scale, WHOQOL questionnaire and FSFI questionnaire at the first visit, 3-month and 6-month follow-up.
  WHOQOL questionnaire (The World Health Organization Quality of life)application for evaluation at the first visit, 3-month and 6-month follow-up.
  FSFI questionnaire application for evaluation of sexual function at the first visit, 3-month and 6-month follow-up.
  Interventions: Behavioral: WHOQOL questionnaire; Behavioral: FSFI questionnaire; Behavioral: kupperman scale; Drug: tamoxifen; Drug: exemestane

INTERVENTIONS:
Behavioral: WHOQOL questionnaire — WHO defines Quality of Life as individuals perception of their position in life in the context of the culture and value systems in which they live and in relation to their goals, expectations, standards and concerns.
  Other Names: The World Health Organization Quality of Life
Behavioral: FSFI questionnaire — FSFI questionnaire application for evaluation of sexual function at the first visit, 3-month and 6-month follow-up.
  Other Names: Female sexual function index (FSFI) questionnaire
Behavioral: kupperman scale — Kupperman scale is a tool to help evaluate the severity of menopausal symptoms
  Other Names: Blatt-Kupperman menopausal index
Drug: Cimicifuga racemosa — The Cimicifuga racemosa effects on the sexuality of women with Breast cancer
  Other Names: Black Cohosh
  Arms: Cimicifuga racemosa
Drug: tamoxifen — The Cimicifuga racemosa effects on the sexuality of women with Breast cancer using tamoxifen
Drug: exemestane — The Cimicifuga racemosa effects on the sexuality of women with Breast cancer using aromatase inhibitor.
  Other Names: aromatase inhibitor

SUMMARY:
The purpose of this study is to evaluate the Cimicifuga racemosa effects on the sexuality of women with Breast cancer using tamoxifen or aromatase inhibitor through questionnaires.

DETAILED DESCRIPTION:
For the study will be recruited 60 women treated with breast cancer, using tamoxifen or aromatase inhibitor, are in menopause, hot flashes and has with or without sexual life. They will answer the questionnaires: Kupperman, World Health Organization Quality of Life (WHOQOL) and those sexually active will have Female Sexual Function Index (FSFI). The control group will have 30 patients using tamoxifen alone or inhibitor. The other group will have 30 patients receiving tamoxifen or inhibitor and will start with 2 tablets per day of dry extract of Cimicifuga racemosa. They will be followed for 6 months and answer questionnaires at the first visit, 3-month and 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Menopausal women with breast cancer treated and using tamoxifen or aromatase inhibitor.
* With hot flashes and with or without active sexual life.

Exclusion Criteria:

* Women did not have breast cancer
* do not use tamoxifen or aromatase inhibitor
* not in menopause and not have hot flashes

Ages: 48 Years to 68 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-09 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Hot flashes (score of hot flashes) | 6 months
  Determine the score of hot flashes

SECONDARY OUTCOMES:
Sexual function (score of sexual function questionnaire (FSFI) | 3 months
  Determine the score of sexual function questionnaire (FSFI)
Sexual function (score of sexual function questionnaire (FSFI) | 6 months
  Determine the score of sexual function questionnaire (FSFI)

OTHER OUTCOMES:
Quality of life (questionnaire scores of quality of life (WHOQOL) | 3 months
  Determine the questionnaire scores of quality of life (WHOQOL)
Quality of life (questionnaire scores of quality of life (WHOQOL) | 6 months
  Determine the questionnaire scores of quality of life (WHOQOL)

CONTACTS AND LOCATIONS:
Overall Officials: Black cohosh, Principal Investigator — Irmandade da Santa Casa Misericordia Sao Paulo
Locations (1):
- Carolina Furtado Macruz, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
When I have finished my recruitment and analysis of the results.